CLINICAL TRIAL: NCT05043246
Title: Safety and Immune Response of COVID-19 Vaccination in Patients With Basic Disease
Acronym: SIM-PBD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Hong Ren, Dr/ Prof., The Second Affiliated Hospital of Chongqing Medical University
Other Study IDs: 2021-49
Record Dates: First submitted 2021-08-12; First posted 2021-09-14 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Diseases, Chronic; Covid19; Adverse Reaction to Vaccine
Keywords: COVID-19; vaccine; basic diseases; cancer diseases
MeSH Terms: conditions — Chronic Disease; COVID-19 | interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Basic diseases Patients/Healthy People: Hypertension, diabetes, chronic obstructive pulmonary disease, chronic kidney disease,Chronic Liver Diseases, Cancer diseases Patients
  Interventions: Biological: SARS-COV-2 VACCINE

INTERVENTIONS:
Biological: SARS-COV-2 VACCINE — the antibody titer and adverse reactions were observed.

SUMMARY:
On 11 February 2020, the International Committee for the Classification of Viruses named the disease caused by SAＲS-CoV-2 infection in humans as the new coronavirus pneumonia (coronavirus disease 2019, COVID-19).Due to the decline of immunity and cardiopulmonary function in patients with basic diseases (hypertension, diabetes, chronic obstructive pulmonary disease, chronic kidney disease, cancer diseases, etc.), COVID-19 's severe illness and mortality mainly increase in these special population. Vaccination of COVID-19 vaccine can effectively prevent COVID-19 virus infection and delay or prevent patients from developing into critical illness and reduce mortality.To evaluate the safety and effectiveness of the population vaccinated with COVID-19 vaccine, and to play a scientific and theoretical supporting role in guiding COVID-19 vaccination scientifically, reasonably and effectively, so this study was carried out.

DETAILED DESCRIPTION:
Due to the decline of immunity and cardiopulmonary function in patients with basic diseases (hypertension, diabetes, chronic obstructive pulmonary disease, chronic kidney disease, cancer diseases, etc.), COVID-19 's severe illness and mortality mainly increase in these special population. At present, there is no evidence that these special population have been vaccinated against COVID-19, but CDC vaccination and the guidelines and consensus of various professional societies hold that: (1) the people with underlying diseases have low immunity and are easy to develop into severe patients with high mortality; (2) although there is no direct evidence of evidence-based medicine, it is best to be vaccinated with COVID-19 vaccine in the absence of disease progression activities to reduce high risk. To evaluate the safety and effectiveness of the population vaccinated with COVID-19 vaccine, and to play a scientific and theoretical supporting role in guiding COVID-19 vaccination scientifically, reasonably and effectively, so this study was carried out.

ELIGIBILITY:
Inclusion Criteria:

* The selection criteria should follow the disease diagnosis guidelines developed by various colleges and the consensus of expert recommendations on vaccination.

Exclusion Criteria:

* The exclusion criteria should follow the disease diagnosis guidelines developed by various colleges and the consensus of expert recommendations on vaccination.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with basic diseases vaccinated with SARS-Cov-2 vaccine.
Sampling Method: Non-Probability Sample
Enrollment: 2300 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events 15 days after vaccination | 15 days：Record the number of adverse reactions such as fever, dizziness, nausea, headache, fatigue, myalgia, etc.
  Evaluate the safety of the vaccine by observing the occurrence of adverse events(such as fever, dizziness, nausea, headache，fatigue, myalgia, etc) and recording the number of subjects with adverse events.
Number of participants with adverse events 30 days after vaccination | 30 days:Record the number of adverse reactions such as fever, dizziness, nausea, headache, fatigue, myalgia, etc.
  Evaluate the safety of the vaccine by observing the occurrence of adverse events(such as fever, dizziness, nausea, headache，fatigue, myalgia, etc) and recording the number of subjects with adverse events.
Number of participants with adverse events 60 days after vaccination | 60 days:Record the number of adverse reactions such as fever, dizziness, nausea, headache, fatigue, myalgia, etc.
  Evaluate the safety of the vaccine by observing the occurrence of adverse events(such as fever, dizziness, nausea, headache，fatigue, myalgia, etc) and recording the number of subjects with adverse events.
Number of participants with adverse events 90 days after vaccination | 90 days:Record the number of adverse reactions such as fever, dizziness, nausea, headache, fatigue, myalgia, etc.
  Evaluate the safety of the vaccine by observing the occurrence of adverse events(such as fever, dizziness, nausea, headache，fatigue, myalgia, etc) and recording the number of subjects with adverse events.
Number of participants with adverse events 180 days after vaccination | 180 days:Record the number of adverse reactions such as fever, dizziness, nausea, headache, fatigue, myalgia, etc.
  Evaluate the safety of the vaccine by observing the occurrence of adverse events(such as fever, dizziness, nausea, headache，fatigue, myalgia, etc) and recording the number of subjects with adverse events.
Titer and duration of COVID-19 antibody production 15 days after vaccination | 15 days:Detect the titer and duration of COVID-19 antibodies in the body.
  The titer and duration of COVID-19 antibody were produced at 15 days, 30 days, 90 days, 180 days after vaccination, so as to clarify whether the level of immune response to COVID-19 vaccine was affected in people with basic disease.
Titer and duration of COVID-19 antibody production 30 days after vaccination | 30 days:Detect the titer and duration of COVID-19 antibodies in the body.
  The titer and duration of COVID-19 antibody were produced at 15 days, 30 days, 90 days, 180 days after vaccination, so as to clarify whether the level of immune response to COVID-19 vaccine was affected in people with basic disease.
Titer and duration of COVID-19 antibody production 60 days after vaccination | 60 days:Detect the titer and duration of COVID-19 antibodies in the body.
  The titer and duration of COVID-19 antibody were produced at 15 days, 30 days, 90 days, 180 days after vaccination, so as to clarify whether the level of immune response to COVID-19 vaccine was affected in people with basic disease.
Titer and duration of COVID-19 antibody production 90 days after vaccination | 90 days:Detect the titer and duration of COVID-19 antibodies in the body.
  The titer and duration of COVID-19 antibody were produced at 15 days, 30 days, 90 days, 180 days after vaccination, so as to clarify whether the level of immune response to COVID-19 vaccine was affected in people with basic disease.
Titer and duration of COVID-19 antibody production180 days after vaccination | 180 days:Detect the titer and duration of COVID-19 antibodies in the body.
  The titer and duration of COVID-19 antibody were produced at 15 days, 30 days, 90 days, 180 days after vaccination, so as to clarify whether the level of immune response to COVID-19 vaccine was affected in people with basic disease.

SECONDARY OUTCOMES:
Study on the immune mechanism related to the production of neutralizing antibodies 15 days after vaccination | 15 days:Detect the levels of B cells and related subgroups, Treg and CTL
  After the entire vaccination process was completed, blood was drawn and samples were collected at four nodes 15 days, 30 days, 90 days, and 180 days for the levels of B cells and related subgroups、Treg and CTL.
Study on the immune mechanism related to the production of neutralizing antibodies 30 days after vaccination | 30 days：Detect the levels of B cells and related subgroups, Treg and CTL
  After the entire vaccination process was completed, blood was drawn and samples were collected at four nodes 15 days, 30 days, 90 days, and 180 days for the levels of B cells and related subgroups、Treg and CTL.
Study on the immune mechanism related to the production of neutralizing antibodies 60 days after vaccination | 60 days：Detect the levels of B cells and related subgroups, Treg and CTL
  After the entire vaccination process was completed, blood was drawn and samples were collected at four nodes 15 days, 30 days, 90 days, and 180 days for the levels of B cells and related subgroups、Treg and CTL.
Study on the immune mechanism related to the production of neutralizing antibodies 90 days after vaccination | 90 days：Detect the levels of B cells and related subgroups, Treg and CTL
  After the entire vaccination process was completed, blood was drawn and samples were collected at four nodes 15 days, 30 days, 90 days, and 180 days for the levels of B cells and related subgroups、Treg and CTL.
Study on the immune mechanism related to the production of neutralizing antibodies 180 days after vaccination | 180 days：Detect the levels of B cells and related subgroups, Treg and CTL
  After the entire vaccination process was completed, blood was drawn and samples were collected at four nodes 15 days, 30 days, 90 days, and 180 days for the levels of B cells and related subgroups、Treg and CTL.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Ren, PH D, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University
Locations (1):
- The second affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang L, Xiang F, Wang D, Guo Q, Deng B, Jiang D, Ren H. The safety and immunogenicity of inactivated COVID-19 vaccine in old pulmonary tuberculosis patients. Eur J Clin Microbiol Infect Dis. 2023 Apr;42(4):503-512. doi: 10.1007/s10096-023-04566-0. Epub 2023 Feb 28. PMID 36849838
- [Derived] Xiang F, Long B, He J, Cheng F, Zhang S, Liu Q, Chen Z, Li H, Chen M, Peng M, Yin W, Liu D, Ren H. Impaired antibody responses were observed in patients with type 2 diabetes mellitus after receiving the inactivated COVID-19 vaccines. Virol J. 2023 Feb 7;20(1):22. doi: 10.1186/s12985-023-01983-7. PMID 36750902
- [Derived] Guo Q, Yang L, Peng R, Gao T, Chu X, Jiang D, Ke D, Ren H. Safety and immunogenicity of inactivated COVID-19 vaccine in patients with metabolic syndrome: A cross-sectional observational study. Front Public Health. 2022 Dec 23;10:1067342. doi: 10.3389/fpubh.2022.1067342. eCollection 2022. PMID 36620297